CLINICAL TRIAL: NCT01637857
Title: Oligo-antigenic Diet in the Treatment of Chronic Anal Fissures. Evidence for a Relationship Between Food Hypersensitivity and Anal Fissures
Brief Title: Oligo-antigenic Diet in the Treatment of Chronic Anal Fissures.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Pasquale Mansueto, MD, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACPM01
Record Dates: First submitted 2012-07-08; First posted 2012-07-11 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Anal Fissures Treatment and Oligoantigenic Diet
Keywords: foof hypersensitivity; anal fissures; ano-rectal manometry
MeSH Terms: conditions — Fissure in Ano

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lifestyle counseling (Sham Comparator): Group of patients treated with sham oligoantigenic diet
  Interventions: Dietary Supplement: sham oligoantigenic diet associated to lifestyle instruction
- oligoantigenic diet (Experimental): Treatment with oligoantigenic diat
  Interventions: Dietary Supplement: oligoantigenic diet

INTERVENTIONS:
Dietary Supplement: sham oligoantigenic diet associated to lifestyle instruction — sham oligoantigenic diet associated to lifestyle instruction
  Arms: lifestyle counseling
Dietary Supplement: oligoantigenic diet — oligoantigenic diet associated to life style counseling
  Arms: oligoantigenic diet

SUMMARY:
Patients with chronic constipation due to food hypersensitivity (FH) had an elevated anal sphincter resting pressure. No studies have investigated a possible role of FH in anal fissures (AF). We aim to evaluate the effectiveness of a diet in curing AF and the clinical effects of a double-blind placebo controlled (DBPC) challenge with cow's milk protein or wheat.

DETAILED DESCRIPTION:
Context: Patients with chronic constipation due to food hypersensitivity (FH) had an elevated anal sphincter resting pressure. No studies have investigated a possible role of FH in anal fissures (AF).

Objective: We aim to evaluate 1) the effectiveness of a diet in curing AF; 2) the clinical effects of a double-blind placebo controlled (DBPC) challenge with cow's milk protein or wheat.

Design: The study will have two different parts: the first to verify the effectiveness of the oligo-antigenic diet in chronic AF treatment; the second to search for a possible cause-effect relationship between the diet and the onset of the AF.

Setting: We will enrol consecutive adult patients with chronic AF who will refer to a Surgical Department of the University of Palermo for a 3-years period. Inclusion criteria are: evidence of CAF evaluated by an experienced rectal surgeon; patient age >16 years. Exclusion criteria are: a diagnosis of inflammatory bowel disease, ongoing steroid treatment performed for any reason, an exclusion diet followed for any reason, and pregnancy. At the time of the first evaluation, routine laboratory tests, immunology tests, rectal biopsies and anal-rectal manometry will be performed.

Patients: patients, finally included in the study, will be randomized to one of the treatment groups.

Interventions: Enrolled patients will be randomized to receive a "true elimination diet" or a "sham elimination diet"; both groups will also receive topical nifedipine and lidocaine.

Main Outcome Measures: The patients will be evaluated every two weeks for CAF persistence or healing; anal pain will be scored on a visual analogue scale ranging from 0 (absence of pain) to 10 (intolerable pain). Anal-rectal manometry will be repeated at the end of the study period, in all patients who will be treated.

ELIGIBILITY:
Inclusion Criteria:

* evidence of chronic anal fissures evaluated by an experienced rectal surgeon
* patient age >16 years.

Exclusion Criteria:

* a diagnosis of inflammatory bowel disease
* ongoing steroid treatment performed for any reason
* an exclusion diet followed for any reason
* pregnancy.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2006-01; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Chronic anal fissures persistence or healing | 2 years
  The patients will be evaluated every two weeks for eight weeks for CAF persistence or healing; anal pain will be scored on a visual analogue scale ranging from 0 (absence of pain) to 10 (intolerable pain). Anal-rectal manometry will be repeated at the end of the study period, in all patients who will be treated.

SECONDARY OUTCOMES:
Anal fissures recurring after Double-Blind Placebo-Controlled food challenge | 2 years
  In this part of the study will be included patients with healed chronic anal fissures on true elimination diet (GROUP B) plus patients of GROUP A, who received "sham elimination diet", uncured, were offered the treatment option of "true elimination diet" before undergoing surgery, accepted, and finally cured. Therefore, we will evaluate anal fissures recurring after Double-Blind Placebo-Controlled Food Challenges with cow's milk and wheat, and Open Challenges with other foods (i.e. egg, tomato and chocolate).

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carroccio, Prof., Study Director — Internal Medicine, Hospital of Sciacca, ASP Agrigento, University of Palermo, Italy; Pasquale Mansueto, Dr., Principal Investigator — University of Palermo; Sebastiano Bonventre, Dr., Principal Investigator — University of Palermo
Locations (1):
- Surgery Department, University of Palermo, Italy, Palermo, Italy, Italy